CLINICAL TRIAL: NCT05282030
Title: An Open-label, Multi-center Phase 1 Pharmacokinetic and Tolerability Study of Tolebrutinib Given as a Single Oral Dose in Participants With Renal Impairment and in Matched Participants With Normal Renal Function.
Brief Title: Study to Assess the Plasma Concentration of Tolebrutinib Given as a Tablet to Adult Participants With Renal Impairment Compared to Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP16399; U1111-1269-6877 (Registry Identifier: ICTRP); POP16399 (Other: Sanofi Identifier); 2021-006685-20 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Severe Renal Impairment (RI) group (Part A only) (Experimental): Single dose of tolebrutinib (SAR442168) will be administered on Day 1 under fed condition
  Interventions: Drug: tolebrutinib
- Normal Renal Function group (Part A and B) (Experimental): Single dose of tolebrutinib (SAR442168) will be administered on Day 1 under fed condition
  Interventions: Drug: tolebrutinib
- Moderate RI group (Part B only conditional) (Experimental): Single dose of tolebrutinib (SAR442168) will be administered on Day 1 under fed condition
  Interventions: Drug: tolebrutinib

INTERVENTIONS:
Drug: tolebrutinib — Pharmaceutical form: Film-coated tablets Route of administration: oral

SUMMARY:
The purpose of this parallel group, Phase 1, open-label, 2-arm study is to assess the effect of severe (Part A) and moderate (Part B, conditional) renal impairment (RI) on pharmacokinetics (PK), safety and tolerability of tolebrutinib tablets compared with normal renal function, in male and female participants aged 18 to 79 years.

DETAILED DESCRIPTION:
The total duration of the study per participant will be up to 38 days including:

* A screening period of up to 4 weeks.
* A 5-day, open-label treatment period.
* Up to 7 days post-treatment follow-up period

ELIGIBILITY:
Inclusion Criteria:

* For participants with severe RI (Part A): Absolute GFR <30 mL/min, and not requiring dialysis (based on estimated glomerular filtration rate [eGFR] by absolute GFR from the MDRD formula with individual BSA, without race correction), with a variability within +/- 20% between screening and Day -1 assessments.
* For participants with moderate RI (Part B conditional): 30 mL/min ≤ absolute GFR ≤59 mL/min (based on estimated glomerular filtration rate [eGFR] by absolute GFR from the MDRD formula with individual body surface area (BSA), without race correction), with a variability within +/- 20% between screening and Day -1 assessments
* For participants with normal renal function: Absolute GFR ≥ 90 mL/min (based on eGFR by absolute GFR from the MDRD formula with individual BSA, without race correction), with a variability within +/- 20% between screening and Day -1 assessments.

For all participants:

* Body weight between 50.0- and 115.0 kg, inclusive, if male, between 40.0 and 100 kg, inclusive, if female, and body mass index (BMI) between 18 to 40 kg/m2 inclusive, at screening.
* Participant with platelet count ≥150 000/μL at the screening visit and at Day -1

Exclusion Criteria:

For all participants:

* Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension, defined as a decrease in SBP≥30 mmHg within 3 minutes when changing from a supine to a standing position at screening and Day -1
* Blood donation (usually approximately 500 mL), within 2 months before inclusion.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* History of alcohol or drug abuse within 1 year prior to screening
* Smoking regularly more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 8 cigarettes per day during the institutionalization.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 72 hours before inclusion
* Use of any herbal medicines 2 weeks before IMP administration
* Treatment with a strong, moderate or mild CYP2C8 inducer or inhibitor, OR a strong, moderate or mild CYP3A inducer, OR a strong, or moderate CYP3A inhibitor, within 14 days before the study treatment administration or 5 half-lives, whichever is longer

Specific criteria for participants with RI

* Active liver disease, cirrhosis, chronic liver disease, hepatic insufficiency
* Acute renal failure (de novo or superimposed to preexisting chronic RI), nephrotic syndrome.
* History of or current hematuria of urologic origin that limits the participant's participation in the study
* Participant requiring dialysis during the study

Specific criteria for participants with normal renal function:

- Any history or presence of clinically relevant hepatic or renal disease

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameters Tolebrutinib: AUC | From Day 1 to Day 4
  Area under the plasma concentration (AUC) versus time curve extrapolated to infinity
Assessment of PK parameters M2: AUC | From Day 1 to Day 4

SECONDARY OUTCOMES:
Assessment of PK parameters Tolebrutinib: Cmax | From Day 1 to Day 4
  Maximum plasma concentration observed (Cmax)
Assessment of PK parameters M2: Cmax | From Day 1 to Day 4
Assessment of PK parameters Tolebrutinib: AUClast | From Day 1 to Day 4
  Area under the serum concentration versus time curve calculated using the trapezoidal method from time zero to the real time AUClast
Assessment of PK parameters M2: AUClast | From Day 1 to Day 4
Number of participants with treatment-emergent adverse events (TEAEs) | From Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (3):
  - Clinical Pharmacology of Miami Site Number : 8400002, Miami, Florida
  - Nucleus Network Site Number : 8400001, Saint Paul, Minnesota
  - Volunteer Research Group-NOCCR Site Number : 8400003, Knoxville, Tennessee
- Investigational Site Number : 2760001, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: POP16399 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25333&tenant=MT_SNY_9011